CLINICAL TRIAL: NCT00513188
Title: A Pilot Study of the Efficacy of the Chop-Montak Regimen in Patients With Newly Diagnosed Peripheral T Cell Lymphoma
Brief Title: Combination Chemotherapy and Denileukin Diftitox in Treating Patients With Newly Diagnosed T-Cell Non-Hodgkin Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 20060912; SCCC-2006068
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; adult nasal type extranodal NK/T-cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Extranodal NK-T-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — denileukin diftitox; Cyclophosphamide; Cytarabine; Doxorubicin; Leucovorin; Methotrexate; Prednisone; Vincristine; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: denileukin diftitox
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: leucovorin calcium
Drug: methotrexate
Drug: prednisone
Drug: vincristine sulfate
Genetic: protein expression analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Combinations of biological substances in denileukin diftitox may be able to carry cancer-killing substances directly to non-Hodgkin lymphoma cells. Giving combination chemotherapy together with denileukin diftitox may kill more cancer cells.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy together with denileukin diftitox works in treating patients with newly diagnosed T-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate failure-free survival of patients with newly diagnosed peripheral T-cell non-Hodgkin lymphoma treated with cyclophosphamide, doxorubicin hydrochloride, vincristine, prednisone (CHOP), and denileukin diftitox (Ontak®) alternating with high-dose methotrexate, leucovorin calcium, cytarabine, and Ontak® (CHOP-MONTAK regimen).

Secondary

* To determine the response rate (CR, CRu, and PR) in these patients.
* To determine the overall survival of these patients.
* To determine the toxicity profile of this regimen.
* To correlate response with CD25 expression in these patients.

OUTLINE:

* Courses 1, 3, and 5: Patients receive cyclophosphamide IV over 30 minutes, doxorubicin hydrochloride IV, and vincristine IV on day 1; oral prednisone once daily on days 1-5; and denileukin diftitox IV over 60 minutes on days 1 and 2. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Courses 2, 4, and 6: Patients receive high-dose methotrexate (MTX) IV over 24 hours on day 1; cytarabine IV over 2 hours every 12 hours on days 2 and 3; and leucovorin calcium IV over 15 minutes every 6 hours for 8 doses beginning 12 hours after the last dose of each MTX infusion. Patients also receive denileukin diftitox IV over 60 minutes for 2 doses once MTX blood levels have cleared. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for correlative studies. Samples are analyzed for CD25-positive or -negative expression and response rate via flow cytometry.

After completion of study treatment, patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of peripheral T-cell non-Hodgkin lymphoma

  * Newly diagnosed, previously untreated disease
  * Mycosis fungoides with systemic disease (i.e., beyond the skin) allowed
* No CD30-positive ALK 1-positive T-anaplastic large cell lymphoma
* No skin only involvement
* No localized NK/T-cell lymphoma
* No adult T-cell leukemia/lymphoma
* No known CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* ANC > 1,000/mm^3 (unless due to lymphoma)
* Platelets > 100,000/mm^3 (unless due to lymphoma)
* Serum bilirubin ≤ 2.0 mg/dL (unless due to lymphoma)
* Serum creatinine ≤ 1.5 mg/dL (unless due to lymphoma)
* Albumin ≥ 3.0 g/dL
* Cardiac ejection fraction ≥ 50% by MUGA or echocardiogram
* Not pregnant or nursing
* Negative serum or urine β-HCG at screening
* Women and male partners of child-bearing potential must practice an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch) before study entry and throughout the study period
* Willing to receive transfusions of blood products
* No HIV-positive serology
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Child's class C liver cirrhosis
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit study compliance
* No other prior or concurrent malignancy with a poor prognosis (i.e., < 90% probability of survival at 5 years) or that is actively being treated

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for the treatment of lymphoma
* No other concurrent investigational agents for the treatment of lymphoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Failure-free survival

SECONDARY OUTCOMES:
Response rate (CR, CRu, and PR)
Overall survival
Toxicity profile
Correlation of response with CD25 expression

CONTACTS AND LOCATIONS:
Overall Officials: Maricer Escalon, MD, MS, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States